CLINICAL TRIAL: NCT06349967
Title: Nab-paclitaxel Combined With Cadonilimab (AK104) for the Second-line Treatment of Advanced Gastric Cancer: A Prospective, Multicenter, Single-arm, Phase II Study
Brief Title: Nab-paclitaxel Combined With Cadonilimab (AK104) for the Second-line Treatment of Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH-2023-1592
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel+Cadonilimab (AK104) (Experimental): Nab-paclitaxel 100mg/m2 ivgtt d1, d8, d15, q28d; Cadonilimab (AK104) 6mg/kg ivgtt d1, d15, q28d;
  Interventions: Drug: Nab-paclitaxel Combined With Cadonilimab (AK104)

INTERVENTIONS:
Drug: Nab-paclitaxel Combined With Cadonilimab (AK104) — Nab-paclitaxel 100mg/m2 ivgtt d1, d8, d15, q28d; Cadonilimab (AK104) 6mg/kg ivgtt d1, d15, q28d;

SUMMARY:
Currently, standard treatment options for gastric cancer failed to first-line treatment include monotherapy with paclitaxel/irinotecan/docetaxel/albumin paclitaxel, or paclitaxel combined with ramucirumab. However, the efficacy of these regimens is still far from satisfactory. The aim of the study is to evaluate the efficacy and safety of nab-paclitaxel combined with cadonilimab for the second-line treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, single arm, phase II clinical study. It is divided into three stages: screening period, treatment period, and follow-up period. The main research objective of this study is to evaluate the objective response rate (ORR) of albumin paclitaxel combined with kandelizumab (AK104) in second-line treatment of gastric cancer with failed first-line fluorouracil/platinum combination immunotherapy. Secondary study objective: To evaluate the disease control rate (DCR), progression free survival (PFS), overall survival (OS), safety, tolerability, and impact on patient quality of life (QoL) of albumin paclitaxel combined with candelizumab (AK104) in second-line treatment of gastric cancer with failed first-line fluorouracil/platinum immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Unresectable gastric/gastroesophageal junction adenocarcinoma diagnosed with peritoneal metastasis through laparoscopic exploration and pathological/cytological examination.
3. No previous antitumor treatment.
4. Agree to provide blood/tissue specimens.
5. The expected survival is longer than 3 months.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status≤1.
7. Adequate organ function including the following:

   1. Total bilirubin ≤1.5 times the upper limit of normal (ULN);
   2. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3×ULN;
   3. Alkaline phosphatase≤2.5×ULN (if the tumor invaded the liver, ≤3×ULN);
   4. Serum creatinine≤1.5×ULN;
   5. Serum amylase and lipase≤1.5×ULN;
   6. International standardized ratio (INR)/partial thromboplastin time (PTT)≤1.5×ULN;
   7. Platelet count ≥ 75,000 /mm3;
   8. Hemoglobin (Hb) ≥ 9 g/dL;
   9. Absolute neutrophil count (ANC) ≥ 1500/mm3;
8. Strict contraception.
9. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Undergoing other clinical trials or having participated in any drug clinical trials one month before enrollment.
2. Hyperprogression occurs in first-line immunotherapy: (1) Tumor burden increased more than 50% compared to baseline upon the first assessment (2-4 cycles of first-line treatment); (2) Tumor growth rate exceeded the previous rate by more than twice after immunotherapy.
3. Active autoimmune disease or history of refractory autoimmune disease.
4. Grade 3-4 immune hepatitis, immune pneumonia, immune myocarditis, etc. appear in first-line immunotherapy.
5. Receiving corticosteroids (>10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding the following therapies: steroid hormone replacement therapy (≤10mg/d); local steroid therapy; and short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting.
6. HER2 positive patients who did not receive trastuzumab in first-line treatment.
7. Active or clinically significant cardiac disease:

   1. Congestive heart failure > New York Heart Association (NYHA) class 2;
   2. Active coronary artery disease;
   3. Arrhythmias requiring treatment other than β-blockers or digoxin;
   4. Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment.
8. Gastrointestinal perforation, obstruction, or uncontrollable diarrhea in the 6 months prior to enrollment.
9. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor was cured and no evidence of disease was found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
10. Patients with a history of HIV infection or active hepatitis B/C.
11. Ongoing > level 2 infection.
12. Symptomatic brain metastasis or meningioma.
13. Unhealed wounds, ulcers or fractures.
14. Renal failure patients requiring blood or peritoneal dialysis.
15. Epileptic that needs medication.
16. Active, symptomatic interstitial lung disease, pleural effusion or ascites that causes breathing difficulties (≥ grade 2 breathing difficulties).
17. History of organ transplantation (including corneal transplantation).
18. Allergy to research drugs or similar drugs, or suspected allergies.
19. Pregnant or lactating women.
20. Medical, psychological or social conditions can affect the recruitment of patients and evaluation of study results.
21. Other antitumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs. Palliative external irradiation for non-target lesions is allowed.
22. Previously used similar chemotherapy drugs or immune checkpoint inhibitors;
23. Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery.
24. Treatment with antitumor Chinese herbal medicine.
25. Vaccination history 4 weeks prior to enrollment
26. The investigator believes that patients who are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | every 3 month postoperation up to 24 months
  the proportion of patients with the best overall response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
disease control rate (DCR) | every 3 month postoperation up to 24 months
  the proportion of patients with the best overall response of CR or PR or stable disease (SD)
overall survival (OS) | every 3 month postoperation up to 24 months
  defined as the time from randomization to death
progression-free survival (PFS) | every 3 month postoperation up to 24 months
  defined as the time from randomization to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Ming Liu, M.D., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei J, Zhang P, Hu Q, Cheng X, Shen C, Chen Z, Zhuang W, Yin Y, Zhang B, Gou H, Yang K, Bi F, Liu M. Nab-paclitaxel combined with cadonilimab (AK104) as second-line treatment for advanced gastric cancer: protocol for a phase II prospective, multicenter, single-arm clinical trial. Front Immunol. 2025 Feb 25;16:1519545. doi: 10.3389/fimmu.2025.1519545. eCollection 2025. PMID 40070819